CLINICAL TRIAL: NCT00154427
Title: A Multi-centre, Randomised, Double-blind, Placebocontrolled, Dose Escalation Trial on Safety and Efficacy of Activated Recombinant Factor VII (rFVIIa/NovoSeven®) in the Treatment of Post-operative Bleeding in Patients Following Cardiac Surgery Requiring Cardiopulmonary Bypass
Brief Title: Use of Activated Recombinant Human Factor VII in Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated after recruiting 172 patients but without proceeding to the highest dosing cohort as this no longer reflects common clinical practice
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7CARD-1610; 2004-000100-40 (EudraCT Number)
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Africa, Asia, Europe, South America and the United States of America (USA).

The trial is planned to investigate the safety and efficacy of NovoSeven® in the management of post-operative bleeding in patients following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative bleeding according to pre-defined criteria for critical bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2004-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Incidence of critical, serious adverse events | Within 30 days

SECONDARY OUTCOMES:
Surgical drainage volume | For the duration of the trial
Amount of transfusions | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (56):
- United States (17):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Camden, New Jersey
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Argentina (5):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Caba
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Corrientes
  - Novo Nordisk Investigational Site, Rosario
- Novo Nordisk Investigational Site, São Paulo, Brazil
- Novo Nordisk Investigational Site, København Ø, Denmark
- France (2):
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Vandœuvre-lès-Nancy
- Germany (8):
  - Novo Nordisk Investigational Site, Aachen
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Cologne
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Krefeld
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Ulm
- India (4):
  - Novo Nordisk Investigational Site, Bangalore
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Trivendrum
- Italy (4):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, San Donato Milanese (MI)
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Singapore, Singapore
- South Africa (3):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (4):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Bilbao
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Seville
- Novo Nordisk Investigational Site, Lund, Sweden
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Southampton

REFERENCES:
- [Result] Gill R, Herbertson M, Vuylsteke A, Olsen PS, von Heymann C, Mythen M, Sellke F, Booth F, Schmidt TA. Safety and efficacy of recombinant activated factor VII: a randomized placebo-controlled trial in the setting of bleeding after cardiac surgery. Circulation. 2009 Jul 7;120(1):21-7. doi: 10.1161/CIRCULATIONAHA.108.834275. Epub 2009 Jun 22. PMID 19546387
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com